CLINICAL TRIAL: NCT02545595
Title: Sugammadex Dosage Based on Ideal Body Weight for Profound Rocuronium-induced Neuromuscular Blockade Reversal in Morbidly Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OBRITI
Record Dates: First submitted 2013-03-27; First posted 2015-09-10 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Morbid Obesity
Keywords: General anaesthesia; Curarization with rocuronium
MeSH Terms: conditions — Obesity, Morbid | interventions — Sugammadex

ARMS (3):
- Sugammadex 1mg/kg (Experimental): for profound rocuronium-induced neuromuscular blockade reversal in morbidly obese patients
  Interventions: Drug: Sugammadex 1 mg/kg
- Sugammadex 2mg/kg (Experimental): for profound rocuronium-induced neuromuscular blockade reversal in morbidly obese patients
  Interventions: Drug: Sugammadex 2 mg/kg
- Sugammadex 4mg/kg (Experimental): for profound rocuronium-induced neuromuscular blockade reversal in morbidly obese patients
  Interventions: Drug: Sugammadex 4 mg/kg

INTERVENTIONS:
Drug: Sugammadex 1 mg/kg
  Arms: Sugammadex 1mg/kg
Drug: Sugammadex 2 mg/kg
  Arms: Sugammadex 2mg/kg
Drug: Sugammadex 4 mg/kg
  Arms: Sugammadex 4mg/kg

SUMMARY:
This randomized double blind clinical trial focuses on patients with Body Masse Index ≥ 40 kg/m2, undergoing scheduled surgery. Neuromuscular transmission monitoring at the adductor is performed using. Anaesthesia is induced with anaesthesic and maintained with curare. At the end of the procedure, patients with profound neuromuscular blockade receive either 1 mg/kg, 2 mg/kg or 4 mg/kg Sugammadex based on ideal body weight. A complete reversal failure is defined by a Train Of Four ratio < 0.9 within 10 min after administration of Sugammadex or if recurarization occurs within 15 min after complete reversal success.

ELIGIBILITY:
Inclusion Criteria:

* General anaesthesia
* Neuromuscular blockade induce by rocuronium
* Body Masse Indice ≥ 40 kg/m2
* informed consent

Exclusion Criteria:

* Contraindication to rocuronium or sugammadex
* Pregnant women
* Severe renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-05; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
determine a profound neuromuscular blockade reversal on ideal body weight | 30 minutes
  A complete reversal failure is defined by a Train Of Four ratio < 0.9 within 10 min after administration of Sugammadex or if recurarization occurs within 15 min after complete reversal success

SECONDARY OUTCOMES:
Compare dosages based on ideal body weight to real body weight | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France